CLINICAL TRIAL: NCT01984359
Title: A Pilot, Single-Center Study Of Quantitative HPV Serum Or Plasma DNA As A Prognostic Marker In P16+/HPV+ Squamous Carcinomas Of The Oropharynx And Unknown Primary Head And Neck Cancers
Brief Title: HPV Serum DNA Levels Predicting Outcome in p16+ Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 22313
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Subjects With p16 Positive/HPV Positive Squamous Cell Carcinomas of the Oropharynx

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): Biosamples will be obtained at multiple time-points for all participants
  Interventions: Other: Obtaining Human tissue

INTERVENTIONS:
Other: Obtaining Human tissue

SUMMARY:
To assess in an exploratory manner, the pronostic utility for locoregional control, progression-free and distant metastasis-free survival of a pre-therapy and post-therapy blood DNA test of HPV E6 and E7 DNA for subtypes 16 and 18 in p16+ and/or HPV+ oropharyngeal cancer patients. This will entail analysis of both initial pre-therapy HPV level as a continuous variable and initial post-therapy HPV level as a dichotomous variable.

ELIGIBILITY:
Inclusion Criteria:

* Histoloically proven primary cancer of the oropharynx, p16(+) and/or HPV (+), who are planned for treatment with resection, radiation and/or chemotherapy.
* Subsites of oropharynx:include tonsil, base of tongue, vallecula, oropharyngeal wall, soft palate, glossotonsillar sulcus.
* No or minimal smoking history (</= 10 pack-year, no smoking in the past 12 months last 10 years based on documented history and/or subject report)
* Age 18 years or older
* Subjects are capable of giving informed consent or have an acceptabl;e surrogate capable of giving consent on the subjects behalf.
* Enrollment on any other study, regardless of therapy is allowed.
* Enrollment on any other tumor or tissue banking study is allowed.
* Patients who have had blood drawn as part of another study, including the IRB-approved ENT Tumor Bank Study, may be included in this study even if the patient has already had surgery.

Exclusion Criteria:

* Previous chemotherapy or radiation therapy to the head and neck unrelated to current disease.
* Previous surgery for head and neck cancer unrelated to current disease.
* Widespread , biopsy-proven metastatic disease (stage IVC disease) at time of presentation (small indeterminate lung or mediastinal nodules are allowed)
* Patients who have started induction chemotherapy prior to consideration for study eligibility.
* Another active cancer except nonmelanomatous skin cancer.
* History of cervical penile or anal cancer.
* Patient treated with surgery, adjuvant radiation therapy or chemotherapy outside of the University of Pennsylvania.
* History of smoking in the past last 12 months 10 years
* History of 10 pack-years of cigarette smoking based on documented history and/or subject report
* Presence of sidespread leukoplakia or erythroplakia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ahn, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States